CLINICAL TRIAL: NCT02106806
Title: Zinc Supplementation on Markers of Oxidative Stress in Post Operative Colorectal Cancer During Chemotherapy Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Selma Freire de Carvalho da Cunha, M.D., PhD, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FAPESP 2011/07867-4
Record Dates: First submitted 2014-03-31; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Chemotherapy; Colorectal Cancer
Keywords: Oxidative stress; Zinc; Chemotherapy; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Zinc; Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Zinc chemotherapy (Experimental): Patients in colorectal chemotherapy supplemented with zinc
  Interventions: Dietary Supplement: Zinc
- Placebo chemotherapy (Placebo Comparator): Patients in colorectal chemotherapy with placebo
  Interventions: Other: Placebo
- Zinc Control (Other): Healthy volunteers supplemented with zinc
  Interventions: Dietary Supplement: Zinc
- Placebo Control (Other): Volunteers received placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc — 35 mg of elemental zinc twice daily for 16 weeks
  Other Names: zinc sulfate
  Arms: Zinc Control; Zinc chemotherapy
Other: Placebo — One capsule, twice daily for 16 weeks
  Other Names: Placebo capsule
  Arms: Placebo Control; Placebo chemotherapy

SUMMARY:
Objective: To determine the oxidative stress during cycles of chemotherapy in patients after surgery for colorectal cancer, with or without oral zinc supplementation. Subjects: Twenty four adults from both genders participated in this study. All patients underwent stage II, III or IV colorectal cancer surgical resection and were starting chemotherapy in HCFMRP- USP. Patients were randomized into two groups. The first one (QTx-Zn Group, n=10) received 70 mg/d of zinc orally and the second one received placebo (QTx-Placebo Group, n=14) for 16 weeks. The study also included 30 healthy volunteers matched for age, gender and socioeconomic status, who received 70 mg/d of zinc supplement (Control-Zn Group, n=21) or placebo (Control-Placebo Group, n=9) for 16 weeks. Methods: The questionnaires about dietary intake (semiquantitative food frequency and food record), fatigue and quality of life (FACIT-F) and questionnaires that assess the side effects of chemotherapy (CTCAE) were evaluated. Anthropometry and bioelectrical impedance measurements were made. Blood collection was performed before the 1st, 2nd, 3rd and 4th cycles of chemotherapy (median duration of 21 days among cicles). Routine laboratory tests, vitamin E and markers anti and pro-oxidants (MDA, SOD, GPx and isoprostane) ere determined. The control group underwent the same procedures, except for chemotherapy. A longitudinal linear mixed effects model was adjusted for each of the variables of interest. The models were fitted using PROC MIXED of SAS version 9 (SAS, CARY, NC, USA). To analyze the association of categorical variables in the different items of the CTCAE, the investigators used the Fisher exact test. Results: The oral zinc supplementation was sufficient to increase plasma levels of zinc and did not alter food intake, body composition and routine laboratory evaluation of patients undergoing chemotherapy for colorectal cancer. Compared with QTx-Placebo Group, QTx-Zn Group showed lower prevalence of complaint on the salivary gland (17 vs. 75%). Fatigue (43 ± 6 vs. 36 ± 13) and quality of life (126 ± 160 vs. 116 ± 27) has become worst in the period between the 1st and 4th cycles of QTx in QTx-Placebo Group. When compared with QTx-Placebo Group, QTx-Zn Group had higher values of SOD before the 1st (2297 ± 503 vs. 1604 ± 352 USOD/g Hb), 2nd (2037 ± 515 vs. 1712 ± 417 USOD/g Hb) and 4th (2202 ± 323 vs. 1821 ± 360 USOD/g Hb) cycles of QTx. GPx values decreased in QTx-Zn Group before the 3rd cycle of QTx (48.5 ± 7.0 vs. 54.3 ± 2.3 mol NADPH/min/gHb). Conclusions: These data suggest that zinc supplementation reduces complaints related to the change in salivary gland, preserving the quality of life and preventing the worsening of fatigue. The increase in SOD can be attributed to zinc supplementation per se, whereas this mineral is a cofactor that endogenous antioxidant enzyme. The highest activity of SOD increases the production of H2O2, whose detoxification involves the participation of GPx, justifying its reduction. There were no changes in plasma levels of vitamin E, MDA and isoprostane during the study period. Considering the values of MDA and isoprostane, the data indicate that regardless of zinc supplementation, the lipid peroxidation of the cell membrane was unchanged during chemotherapy.

DETAILED DESCRIPTION:
Objective: To determine the oxidative stress during cycles of chemotherapy in patients after surgery for colorectal cancer, with or without oral zinc supplementation. Subjects: Twenty four adults from both genders participated in this study. All patients underwent stage II, III or IV colorectal cancer surgical resection and were starting chemotherapy in HCFMRP- USP. Patients were randomized into two groups. The first one (QTx-Zn Group, n=10) received 70 mg/d of zinc orally and the second one received placebo (QTx-Placebo Group, n=14) for 16 weeks. The study also included 30 healthy volunteers matched for age, gender and socioeconomic status, who received 70 mg/d of zinc supplement (Control-Zn Group, n=21) or placebo (Control-Placebo Group, n=9) for 16 weeks. Methods: The questionnaires about dietary intake (semiquantitative food frequency and food record), fatigue and quality of life (FACIT-F) and questionnaires that assess the side effects of chemotherapy (CTCAE) were evaluated. Anthropometry and bioelectrical impedance measurements were made. Blood collection was performed before the 1st, 2nd, 3rd and 4th cycles of chemotherapy (median duration of 21 days among cicles). Routine laboratory tests, vitamin E and markers anti and pro-oxidants (MDA, SOD, GPx and isoprostane) ere determined. The control group underwent the same procedures, except for chemotherapy. A longitudinal linear mixed effects model was adjusted for each of the variables of interest. The models were fitted using PROC MIXED of SAS version 9 (SAS, CARY, NC, USA). To analyze the association of categorical variables in the different items of the CTCAE, the investigators used the Fisher exact test. Results: The oral zinc supplementation was sufficient to increase plasma levels of zinc and did not alter food intake, body composition and routine laboratory evaluation of patients undergoing chemotherapy for colorectal cancer. Compared with QTx-Placebo Group, QTx-Zn Group showed lower prevalence of complaint on the salivary gland (17 vs. 75%). Fatigue (43 ± 6 vs. 36 ± 13) and quality of life (126 ± 160 vs. 116 ± 27) has become worst in the period between the 1st and 4th cycles of QTx in QTx-Placebo Group. When compared with QTx-Placebo Group, QTx-Zn Group had higher values of SOD before the 1st (2297 ± 503 vs. 1604 ± 352 USOD/g Hb), 2nd (2037 ± 515 vs. 1712 ± 417 USOD/g Hb) and 4th (2202 ± 323 vs. 1821 ± 360 USOD/g Hb) cycles of QTx. GPx values decreased in QTx-Zn Group before the 3rd cycle of QTx (48.5 ± 7.0 vs. 54.3 ± 2.3 mol NADPH/min/gHb). Conclusions: These data suggest that zinc supplementation reduces complaints related to the change in salivary gland, preserving the quality of life and preventing the worsening of fatigue. The increase in SOD can be attributed to zinc supplementation per se, whereas this mineral is a cofactor that endogenous antioxidant enzyme. The highest activity of SOD increases the production of H2O2, whose detoxification involves the participation of GPx, justifying its reduction. There were no changes in plasma levels of vitamin E, MDA and isoprostane during the study period. Considering the values of MDA and isoprostane, the data indicate that regardless of zinc supplementation, the lipid peroxidation of the cell membrane was unchanged during chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* colon or rectum adenocarcinoma stages II, III, or IV

Exclusion Criteria:

* liver, kidney, or chronic inflammatory autoimmune diseases;
* active infectious diseases;
* undergoing therapy with immunosuppressant;
* use vitamin or mineral supplementation;
* had been under chemo- or radiotherapy in the previous twelve months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
oxidative stress markers | 18 months
  SOD, GPx, MDA, Isoprostane, Vitamin C, Vitamin E

SECONDARY OUTCOMES:
FACIT-F | 18 months

OTHER OUTCOMES:
CTCAE | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Miranda Ribeiro, R.D., MSc, Principal Investigator — University of Sao Paulo; Selma Freire Cunha, M.D., PhD, Study Director — University of Sao Paulo
Locations (1):
- Division of Medical Nutrition, Department of Internal Medicine, Ribeirão Preto, São Paulo, Brazil